CLINICAL TRIAL: NCT00619385
Title: A Safety and Pharmacokinetic Study of 100 mg, 150 mg and 200 mg of Proellex® Taken for Seven Days by Healthy Adult Female Subjects
Brief Title: A Safety and Pharmacokinetic Study of Proellex®
Acronym: PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZP-003
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Pharmacokinetics
MeSH Terms: interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Proellex 100 mg (Experimental): Proellex 100 mg daily for 7 days
  Interventions: Drug: Proellex
- Proellex 150 mg (Experimental): Proellex 150 mg daily for 7 days
  Interventions: Drug: Proellex
- Proellex 200 mg (Experimental): Proellex 200 mg daily for 7 days
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Proellex — Proellex 25 mg capsules 100 mg, 150 mg or 200mg daily for 7 days
  Other Names: Telapristone acetate

SUMMARY:
Dose escalating study of 7 daily doses of Proellex at 100 mg, 150 mg and 200 mg

DETAILED DESCRIPTION:
This is an open-label, single-center, outpatient, unblinded, multi-dose study of the safety and pharmacokinetic properties of Proellex®. Six female subjects will each receive seven daily doses of Proellex® in separate, rising doses. Dosing must be accomplished between menstrual periods. The first six women will complete the 100 mg visit schedule before the next six women will begin the 150 mg visit schedule. Blood will be collected at pre-dose, and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 5, 8, 12, 24 and 36 (Day 7 only) hrs post-dose on Day 1 and Day 7. Subjects will be allowed to leave the clinic between the 12 and 24 hr and the 24 and 36 hr PK blood draws. Subjects will be discharged from the study after a one month follow-up visit. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to speak, read and understand English and be willing and able to provide written informed consent on an Institutional Review Board (IRB)-approved form prior to the initiation of any study procedures. Subject must have signed and dated a written Informed Consent Form (ICF) before undergoing any study related activities, including discontinuation of any prohibited medications
* Premenopausal women aged 18 - 34 inclusive with body mass index between 18 and 35 inclusive
* Women of child-bearing potential must be willing to use effective non-hormonal, double-barrier method contraception during the study period and for a minimum of 30 days after discontinuation of the study medication. Women who have had a hysterectomy will be allowed into the study
* Must have a negative urine pregnancy test at screening
* Able to swallow gelatin capsules
* In general good health
* Must have agreed to not attempt to become pregnant at any time during study participation or for 30 days thereafter
* Must not have used tobacco (nicotine products) for at least two years before the study starts
* Must have normal (or abnormal and clinically insignificant) laboratory values at screening
* Willing to remain in the clinic for the screening visit and for the treatment visits
* Available for all treatment and follow-up visits
* Willing to comply with all study procedures
* Additional inclusion criteria may apply

Exclusion Criteria:

* Pregnant or lactating females or women who are attempting or expecting to become pregnant at any time during the study
* Past or present history of experiencing any allergic reaction to the formulations administered in this study, or in the opinion of the Principal Investigator, suggests an increased potential for an adverse hypersensitivity
* Any medical condition, which, in the judgment of the Principal Investigator, will prevent the subject from starting and/or completing the study
* Past or present history of any significant cardiovascular, renal, hepatic disease, thrombophlebitis, thromboembolic disorders, or cerebrovascular accident requiring ongoing medical therapy or clinical intervention
* A QTc interval of >450ms at screening
* Subject with abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Principal Investigator
* Subjects with symptomatic uterine fibroids or endometriosis
* Use of other oral contraceptives or hormonal treatments within 30 days of first dose of study medication
* Use of a hormone-releasing intrauterine device
* Subject with a history of alcohol and/or drug abuse
* Known active infection of HIV, Hepatitis A, B or C
* Subject who has participated in a clinical trial with investigational medication within 30 days prior to study medication administration or who plans to take an experimental drug prior to the end of 30 days after participation in this study

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (1):
- Healthcare Discoveries Inc., San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proellex 100 mg | Proellex 150 mg | Proellex 200 mg
Started | 7 | 8 | 10
Completed | 6 | 6 | 6
Not Completed | 1 | 2 | 4
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Other | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proellex 100 mg | Proellex 150 mg | Proellex 200 mg | Total
Number analyzed (Participants) | 7 | 8 | 10 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 10 | 25
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 10 | 25
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Cmax Post Final Dose
Description: To determine the safety and PK properties of 100 mg, 150 mg and 200 mg of Proellex® taken for seven days by healthy adult female subjects.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Proellex 200 mg Caps: Proellex 200 mg daily for 7 days capsules
- Proellex 200 mg Vials: Proellex 200 mg daily for 7 days vials
Arm/Group | Proellex 100 mg | Proellex 150 mg | Proellex 200 mg Caps | Proellex 200 mg Vials
Number analyzed (Participants) | 6 | 6 | 3 | 3
ng/mL | 1944 (625) | 3807 (1670) | 2293 (1319) | 2777 (954)

2. Primary Outcome: AUC Post Final Dose
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Groups:
- Proellex 200 mg Caps: Proellex 200 mg capsules daily for 7 days
- Proellex 200 mg Vials: Proellex 200 mg vials daily for 7 days
Arm/Group | Proellex 100 mg | Proellex 150 mg | Proellex 200 mg Caps | Proellex 200 mg Vials
Number analyzed (Participants) | 6 | 6 | 3 | 3
hour*ng/mL | 57591 (70514) | 137634 (146024) | 230731 (371463) | 190324 (95387)

ADVERSE EVENTS:
Arm/Group | Proellex 100 mg | Proellex 150 mg | Proellex 200 mg
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 6/7 | 6/8 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proellex 100 mg (N=7) | Proellex 150 mg (N=8) | Proellex 200 mg (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
UTI (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginitis trichomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Amenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Oligomenorrhea (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights